CLINICAL TRIAL: NCT02787395
Title: Patients Education of a Self-reduction Technique for Anterior Dislocation of Shoulder
Brief Title: Self Reduction of Shoulder Dislocation
Acronym: SR-SD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-15-OC-0612-CTIL
Record Dates: First submitted 2016-05-22; First posted 2016-06-01 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Anterior Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milch (Experimental): modified Milch technique for self reduction
  Interventions: Procedure: shoulder dislocation self reduction
- Boss Holtzach (Experimental): Boss Holtzach technique for self reduction
  Interventions: Procedure: shoulder dislocation self reduction
- Stimson (Experimental): Stimson technique for self reduction
  Interventions: Procedure: shoulder dislocation self reduction

INTERVENTIONS:
Procedure: shoulder dislocation self reduction — shoulder dislocation self reduction using one of three methods in the study

SUMMARY:
Anterior dislocation of the shoulder (glenohumeral joint) is one of the most prevalent dislocations. Following a first dislocation recurrence rates of up to 80% have been reported. Many patients will seek medical assistance for reduction of the shoulder after each of these recurrent dislocations. The investigators describe the results of reduction of anterior glenohumeral dislocation using a modified self manipulated Milch technique that can be performed by the patients themselves after simple guidance and demonstration. This method is directed to patients who are not willing or cannot have surgical stabilization and may be in a place where medical assistance is not available.

ELIGIBILITY:
Inclusion Criteria:

* anterior shoulder dislocation
* acute (24 hours) shoulder dislocation

Exclusion Criteria:

* shoulder fracture
* non-cooperative patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
rate of successfull self reduction | 10 minutes
  the number/rate of successful reductions using each technique will be calculated

SECONDARY OUTCOMES:
pain using VAS during reduction | 10 minutes
  patients will be asked to report pain levels using VAS during the self reduction procedure
patient satisfaction from self reduction process using VAS | 10 minutes
  patients will be asked to report their satisfaction from self reduction process using VAS

IPD SHARING:
Plan to Share IPD: No